CLINICAL TRIAL: NCT01745952
Title: Multimodal Image-guided Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Refractory Partial Epilepsy.
Brief Title: Treatment of Difficult to Control Focal Epilepsy With Repetitive Transcranial Magnetic Stimulation (rTMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: s52486
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Epilepsies, Partial
Keywords: Epilepsies, Partial; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- figure-of-eight active rTMS coil (Experimental): rTMS is administered using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  Interventions: Device: figure-of-eight active rTMS coil
- round active rTMS coil (Experimental): rTMS is administered using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  Interventions: Device: round active rTMS coil
- sham rTMS coil (figure-of-eight) (Sham Comparator): rTMS is administered using the figure-of-eight sham coil, over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  Interventions: Device: sham rTMS coil (figure-of-eight)

INTERVENTIONS:
Device: figure-of-eight active rTMS coil — navigated rTMS over epileptogenic focus using figure-of-eight active rTMS coil
  Arms: figure-of-eight active rTMS coil
Device: round active rTMS coil — navigated rTMS over epileptogenic focus using round active rTMS coil
  Arms: round active rTMS coil
Device: sham rTMS coil (figure-of-eight) — commercially available placebo coil that provides slight sensory stimulation and discharge noise without stimulating cortical tissue
  Arms: sham rTMS coil (figure-of-eight)

SUMMARY:
The investigators will treat patients with fully characterized refractory unifocal neocortical epilepsy with a technique that delivers magnetic waves (transcranial magnetic stimulation, TMS) to the region that causes the epilepsy. Active rTMS applied over the epileptogenic focus will reduce seizure frequency compared with sham rTMS.

DETAILED DESCRIPTION:
1. Background and study aims

   Epilepsy is a disease that causes repetitive seizures. In 60% of people with epilepsy, these seizures start in a small zone of the brain (focal or partial epilepsy). This zone can be in the depth of the temporal lobe (mesial temporal lobe epilepsy) or in another brain region (neocortical epilepsy). Even with optimal medical care, up to 30% of people with epilepsy continue to have seizures.

   The investigators will treat people with neocortical partial epilepsy with a technique that delivers magnetic waves (transcranial magnetic stimulation, TMS) to the region that causes the epilepsy. The investigators have good reasons to believe that there will be fewer seizures during several weeks after treatment.
2. Who can participate?

   You have neocortical focal epilepsy. A doctor who specializes in epilepsy made this diagnosis. You had at least one seizure recorded while in an epilepsy monitoring unit. You had an MRI scan of the brain. You can deliver us all the results of the tests you had.

   You continue to have more than 4 seizures a month. You tried a least two different schemes of anti-epileptic drugs as prescribed by your doctor and those schemes were well tolerated. Nevertheless this never cured the seizures.

   You are older than 16 years. You don't plan to become pregnant during the study. You need to faithfully continue your treatment as prescribed by your doctor and don't change the drugs you take from at least 4 weeks before the study until 8 weeks after the last TMS session. You need to be able to keep a diary of your seizures.
3. What does the study involve?

   You will need to come to the hospital every weekday during two consecutive weeks, every three months during nine months for the TMS-treatment. So you will have three treatment sessions. You will have a brain scan (FDG-PET) before the first treatment and after each session.

   The magnetic pulses will be delivered differently during each of the three treatment sessions: once on a rather small area of the brain, once on a larger brain area and once using a dummy coil, i.e. you will have two active treatment sessions and one dummy or placebo session. The investigators will not tell in which order they deliver the treatments.
4. What are the possible benefits and risks of participating?

The investigators have good reasons to believe you will have fewer seizures in the weeks following the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* fully characterized refractory unifocal neocortical epilepsy (i.e. the epileptogenic zone is well defined)
* on a stable drug regimen for at least one month,
* able to complete a seizure dairy either by the patient or by a significant other

Exclusion Criteria:

* Metal in the head including deep brain stimulators, aneurysmal clips, ventricular shunts, cochlear implants, ossicular reconstruction of the middle ear…
* pacemaker, implantable cardioverter-defibrillator (ICD)
* psychogenic non-epileptic seizures and other non-epileptic spells

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Van Paesschen Wim, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, department of Neurology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun W, Mao W, Meng X, Wang D, Qiao L, Tao W, Li L, Jia X, Han C, Fu M, Tong X, Wu X, Wang Y. Low-frequency repetitive transcranial magnetic stimulation for the treatment of refractory partial epilepsy: a controlled clinical study. Epilepsia. 2012 Oct;53(10):1782-9. doi: 10.1111/j.1528-1167.2012.03626.x. Epub 2012 Sep 5. PMID 22950513
- [Background] Fregni F, Otachi PT, Do Valle A, Boggio PS, Thut G, Rigonatti SP, Pascual-Leone A, Valente KD. A randomized clinical trial of repetitive transcranial magnetic stimulation in patients with refractory epilepsy. Ann Neurol. 2006 Oct;60(4):447-55. doi: 10.1002/ana.20950. PMID 17068786
- [Background] Theodore WH, Hunter K, Chen R, Vega-Bermudez F, Boroojerdi B, Reeves-Tyer P, Werhahn K, Kelley KR, Cohen L. Transcranial magnetic stimulation for the treatment of seizures: a controlled study. Neurology. 2002 Aug 27;59(4):560-2. doi: 10.1212/wnl.59.4.560. PMID 12196649
- [Background] Cantello R, Rossi S, Varrasi C, Ulivelli M, Civardi C, Bartalini S, Vatti G, Cincotta M, Borgheresi A, Zaccara G, Quartarone A, Crupi D, Lagana A, Inghilleri M, Giallonardo AT, Berardelli A, Pacifici L, Ferreri F, Tombini M, Gilio F, Quarato P, Conte A, Manganotti P, Bongiovanni LG, Monaco F, Ferrante D, Rossini PM. Slow repetitive TMS for drug-resistant epilepsy: clinical and EEG findings of a placebo-controlled trial. Epilepsia. 2007 Feb;48(2):366-74. doi: 10.1111/j.1528-1167.2006.00938.x. PMID 17295632
- [Background] Tergau F, Naumann U, Paulus W, Steinhoff BJ. Low-frequency repetitive transcranial magnetic stimulation improves intractable epilepsy. Lancet. 1999 Jun 26;353(9171):2209. doi: 10.1016/S0140-6736(99)01301-X. No abstract available. PMID 10392988
- [Background] Daniele O, Brighina F, Piazza A, Giglia G, Scalia S, Fierro B. Low-frequency transcranial magnetic stimulation in patients with cortical dysplasia - a preliminary study. J Neurol. 2003 Jun;250(6):761-2. doi: 10.1007/s00415-003-1080-6. No abstract available. PMID 12862035
- [Background] Tergau F, Neumann D, Rosenow F, Nitsche MA, Paulus W, Steinhoff B. Can epilepsies be improved by repetitive transcranial magnetic stimulation?--interim analysis of a controlled study. Suppl Clin Neurophysiol. 2003;56:400-5. doi: 10.1016/s1567-424x(09)70244-2. No abstract available. PMID 14677417
- [Background] Brasil-Neto JP, de Araujo DP, Teixeira WA, Araujo VP, Boechat-Barros R. Experimental therapy of epilepsy with transcranial magnetic stimulation: lack of additional benefit with prolonged treatment. Arq Neuropsiquiatr. 2004 Mar;62(1):21-5. doi: 10.1590/s0004-282x2004000100004. Epub 2004 Apr 28. PMID 15122428
- [Background] Kinoshita M, Ikeda A, Begum T, Yamamoto J, Hitomi T, Shibasaki H. Low-frequency repetitive transcranial magnetic stimulation for seizure suppression in patients with extratemporal lobe epilepsy-a pilot study. Seizure. 2005 Sep;14(6):387-92. doi: 10.1016/j.seizure.2005.05.002. PMID 16046153
- [Background] Santiago-Rodriguez E, Cardenas-Morales L, Harmony T, Fernandez-Bouzas A, Porras-Kattz E, Hernandez A. Repetitive transcranial magnetic stimulation decreases the number of seizures in patients with focal neocortical epilepsy. Seizure. 2008 Dec;17(8):677-83. doi: 10.1016/j.seizure.2008.04.005. Epub 2008 May 20. PMID 18495500
- [Background] Joo EY, Han SJ, Chung SH, Cho JW, Seo DW, Hong SB. Antiepileptic effects of low-frequency repetitive transcranial magnetic stimulation by different stimulation durations and locations. Clin Neurophysiol. 2007 Mar;118(3):702-8. doi: 10.1016/j.clinph.2006.11.008. Epub 2007 Jan 16. PMID 17223384
- [Result] Seynaeve L, Devroye A, Dupont P, Van Paesschen W. Randomized crossover sham-controlled clinical trial of targeted low-frequency transcranial magnetic stimulation comparing a figure-8 and a round coil to treat refractory neocortical epilepsy. Epilepsia. 2016 Jan;57(1):141-50. doi: 10.1111/epi.13247. Epub 2015 Dec 8. PMID 26642974
- [Result] Seynaeve L, Van Paesschen W. Response to "Safety of repetitive transcranial magnetic stimulation in patients with epilepsy: A systematic review" by Luisa Santos Pereira and colleagues. Epilepsy Behav. 2016 Sep;62:308. doi: 10.1016/j.yebeh.2016.07.002. Epub 2016 Aug 1. No abstract available. PMID 27492628

RESULTS

PARTICIPANT FLOW:
Groups:
- Figure-of-eight Active Coil; Then Round Active Coil; Then Sham: * rTMS using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the sham coil, over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
- Round Active Coil; Then Sham; Then Figure-of-eight Active Coil: * rTMS using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the sham coil, over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
- Sham Coil; Then Figure-of-eight Active Coil; Then Round Active: * rTMS using the sham coil over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the figure-of-eight active coil, at 90% of the resting motor threshold, over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
  * rTMS using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  * 12 week follow-up period
Period: Overall Study
Arm/Group | Figure-of-eight Active Coil; Then Round Active Coil; Then Sham | Round Active Coil; Then Sham; Then Figure-of-eight Active Coil | Sham Coil; Then Figure-of-eight Active Coil; Then Round Active
Started | 4 | 4 | 3
Completed | 3 | 3 (data of one patient not used due to no seizure diary entries on multiple occasions) | 3
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: description of the patients at the onset of the study
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [24 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
baseline seizure frequency per week [Mean (Full Range); unit: seizures/week] | 24.9 [0.5 to 124.6]

OUTCOME MEASURES:

1. Primary Outcome: 50% Responder Rate After Active rTMS Treatment Compared With Placebo Treatment
Description: Number of participants achieving a 50% or greater reduction in seizure frequency from baseline
Time Frame: week 12 after each intervention
Population: Besides the reported participants that went through whole protocol, one supplementary participant underwent the first rTMS session of the first protocol and one supplementary participant underwent the first rTMS session of the second protocol
Measure: Number; unit: participants
Arm/Group | Figure-of-eight Active Coil; Then Round Active Coil; Then Sham | Round Active Coil; Then Sham; Then Figure-of-eight Active Coil | Sham Coil; Then Figure-of-eight Active Coil; Then Round Active
Number analyzed (Participants) | 3 | 2 | 3
participants
  50% seizure reduction over any of three periods | 0 | 0 | 0
  50% seizure reduction over whole study | 0 | 0 | 0

2. Secondary Outcome: Seizure Frequency After Active rTMS Treatment Compared With Placebo Treatment
Description: Seizure frequency was recorded in patient diaries and reviewed with the neurologist/epileptologist (outcomes assessor) at visits 12 weeks (+/- 1 week) after each intervention. The average weekly seizure rate was calculated and compared to baseline frequency over all participants.
Time Frame: week 12 after each treatment
Population: baseline weekly seizure frequency over all participants was 24.8 (95% confidence interval 8.2-76.1)
Measure: Mean (95% Confidence Interval); unit: seizures/week
Groups:
- Figure-of-eight Active rTMS Coil: rTMS is administered using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  All patients who have undergone this treatment are taken together, irrespective of order the other treatments were administered.
- Round Active rTMS Coil: rTMS is administered using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  All patients who have undergone this treatment are taken together, irrespective of order the other treatments were administered
- Sham rTMS Coil (Figure-of-eight): rTMS is administered using the figure-of-eight sham coil, over the epileptogenic region, in trains of 500 pulses with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  All patients who have undergone this treatment are taken together, irrespective of order the other treatments were administered
Arm/Group | Figure-of-eight Active rTMS Coil | Round Active rTMS Coil | Sham rTMS Coil (Figure-of-eight)
Number analyzed (Participants) | 8 | 9 | 7
seizures/week | 25.7 [7.4 to 89.4] | 23.5 [7.2 to 76.2] | 28.6 [8.2 to 99.8]

3. Other Pre Specified Outcome: Alteration of Brain Activation as Measured by 18-2-fluoro-2-deoxy-D-glucose Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) on Individual Patient Level
Description: Alterations were assessed by visual inspection of PET scans generated by subtracting the baseline individual PET scan from each of the follow-up scans. The subtraction PET scans were overlayed on the anatomical MRI of the patient and the focus of stimulation determined and an sphere with a 1cm radius around this point was analysed.
Time Frame: within one week after the last treatment day of each session
Population: patients of whom seizure journals were incomplete also included (one participant who went through all 3 trials and one patient of whom journals were not available from the sham session, that was reported by the patient as "ineffective")
Measure: Number; unit: participants
Arm/Group | Figure-of-eight Active rTMS Coil | Round Active rTMS Coil | Sham rTMS Coil (Figure-of-eight)
Number analyzed (Participants) | 9 | 10 | 9
participants
  hypermetabolism compared to baseline | 1 | 3 | 2
  hypometabolism compared to baseline | 3 | 3 | 3

4. Other Pre Specified Outcome: Difference in Seizure Reduction Using Different Coil Types
Description: any difference between the four conditions (baseline/ figure-of-eight treatment/ round coil treatment/ sham treatment) based in negative binomial model for count data
Time Frame: 9 months
Population: averaged weekly seizure count per condition is given for all patients combined
Measure: Mean (95% Confidence Interval); unit: number of seizures per week
Groups:
- Any Difference Between the Four Conditions: effect of baseline/ figure-of-eight/ round/ sham treatment period on the seizure frequency of the patients
Arm/Group | Any Difference Between the Four Conditions
Number analyzed (Participants) | 10
number of seizures per week
  seizures in condition 1 (baseline) | 25 [8 to 76]
  seizures in condition 2 (figure-8) | 26 [7 to 89]
  seizures in condition 3 (round) | 24 [7 to 76]
  seizures in condition 4 (sham) | 29 [8 to 100]
Statistical Analysis 1: Comparison: Any Difference Between the Four Conditions; Test type: Superiority or Other; p = 0.9819, negative binomial model + overdispersion

5. Other Pre Specified Outcome: Questionnaires: Quality of Life in Epilepsy (QOLIE-31), Global Impression of Change-scales, Visual Analogue Scale, Columbia Suicide Severity Rating Scale
Description: * Quality of life in epilepsy (QOLIE-31): self-report (if cognitive faculties allowed) questionnaire of emotional well-being, social functioning, energy/ fatigue, cognitive functioning, seizure worry, medication effects & overall quality of life. Range 0-100, with higher numbers indicating better quality of life.
  * Global impression of change-scales (score 1-7, with 4 no change and lower/higher numbers implying grade of improvement/worsening) and Visual analogue scale (0-10: no problem to horrible): self-report or parent report about effect of treatment
  * Columbia Suicide Severity Rating Scale (CSSR): structured interview about suicidal risk
  * change in QOLIE scores considered better/worse are based on cut-off reported in "DOI 10.1016/j.yebeh.2011.12.023" For global impression of change, the scoring was <4, 4 or >4.
Time Frame: before the first treatment of each session and at the last evaluation visit
Population: * Self-reporting questionnaires could only be filled in by 7 participants For global impression of change scales, the score reached by consensus between the patient and caregiver(s) was used if patient was unable to fill in questionaires: for the three arms, we thus have 7/8/6 scores for each arm respectively
Measure: Number; unit: participants
Arm/Group | Figure-of-eight Active rTMS Coil | Round Active rTMS Coil | Sham rTMS Coil (Figure-of-eight)
Number analyzed (Participants) | 5 | 6 | 5
participants
  better QOLIE score | 3 | 3 | 1
  worse QOLIE score | 0 | 1 | 1
  Global impression of change: no change | 4 | 5 | 5
  Global impression of change: worse | 1 | 1 | 1
  Global impression of change: better | 1 | 1 | 0
  Global impression change: first better, then worse | 1 | 1 | 0
  CSSR-scale increased suicidality | 0 | 0 | 0

6. Other Pre Specified Outcome: Drop Out-rate
Description: exclusion by investigator was due to necessity to change drug regimen due to toxicity
Time Frame: during the 9 months of the study
Population: for this analysis, all patients randomised were included; this includes one patient in the second arm that was not included in any of the other outcome measures, due to lack of reliable outcome parameters
Measure: Number; unit: participants
Arm/Group | Figure-of-eight Active Coil; Then Round Active Coil; Then Sham | Round Active Coil; Then Sham; Then Figure-of-eight Active Coil | Sham Coil; Then Figure-of-eight Active Coil; Then Round Active
Number analyzed (Participants) | 4 | 4 | 3
participants
  excluded by investigator from concluding study | 0 | 1 | 0
  stopped due to intolerance/ inefficiency | 0 | 1 | 0
  stopped due to seizure worsening | 1 | 0 | 0

7. Other Pre Specified Outcome: Adverse Event Rate
Time Frame: during the 9 months of the study
Measure: Number; unit: participants
Arm/Group | Figure-of-eight Active rTMS Coil | Round Active rTMS Coil | Sham rTMS Coil (Figure-of-eight)
Number analyzed (Participants) | 9 | 10 | 8
participants
  worsening seizures | 2 | 1 | 0
  hearing problems | 1 | 1 | 0
  fatigue | 2 | 2 | 2
  concentration difficulties | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 9-month study duration
Groups:
- Figure-of-eight Active rTMS Coil: rTMS is administered using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, at 0.5 Hertz with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  figure-of-eight active rTMS coil: navigated rTMS over epileptogenic focus using figure-of-eight active rTMS coil
- Round Active rTMS Coil: rTMS is administered using the round active coil, at 90% of the resting motor threshold over the epileptogenic region, at 0.5 Hertz with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  round active rTMS coil: navigated rTMS over epileptogenic focus using round active rTMS coil
- Sham rTMS Coil (Figure-of-eight): rTMS is administered using the figure-of-eight sham coil, over the epileptogenic region, at 0.5 Hertz with a total of 1500 pulses per day, during weekdays on two consecutive weeks.
  sham rTMS coil (figure-of-eight): placebo coil that provides slight sensory stimulation and discharge noise without stimulating cortical tissue
Arm/Group | Figure-of-eight Active rTMS Coil | Round Active rTMS Coil | Sham rTMS Coil (Figure-of-eight)
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 3/10 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figure-of-eight Active rTMS Coil (N=9) | Round Active rTMS Coil (N=10) | Sham rTMS Coil (Figure-of-eight) (N=9)
seizure excacerbation (Nervous system disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figure-of-eight Active rTMS Coil (N=9) | Round Active rTMS Coil (N=10) | Sham rTMS Coil (Figure-of-eight) (N=9)
fatigue, concentration difficulties (Nervous system disorders) | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No